CLINICAL TRIAL: NCT03610035
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of NPT189 in Healthy Subjects
Brief Title: A Study of NPT189 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proclara Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPT189-CL001
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2018-12

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Immunoglobulin G

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): NPT189
  Interventions: Drug: NPT189
- Placebo Comparator (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NPT189 — IgG1 Fc-GAIM fusion protein, a recombinant fusion protein
  Other Names: IgG1 (Immunoglobulin G); Fusion Protein; GAIM (General Amyloid Interaction Motif)
  Arms: Experimental
Drug: Placebo — Placebo
  Arms: Placebo Comparator

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of single dose of NPT189 in healthy volunteers. The study will also evaluate the pharmacokinetic characteristics of NPT189.

DETAILED DESCRIPTION:
This study is a Phase1, randomized, double-blind, placebo-controlled, single dose, dose escalation safety and tolerability study of NPT189 in health subjects. Six dose cohorts are planned each with a maximum of 8 participants per cohort. Participants will receive NPT189 by intravenous (IV) or a matching placebo by intravenous infusion. Safety, tolerability, and pharmacokinetics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 and 65 years (inclusive);
* Has provided written informed consent to participate in the study;
* Weigh ≥ 45kg and ≤ 120kg with Body Mass Index of 18-32 inclusive;
* Subject Rescreening: This study does not permit the re-enrollment of a subject who has discontinued from the study as a pre-treatment failure without approval from the sponsor unless the reason they were not included was because the required number of subjects needed at the time of randomization had already been met. Rescreened subjects must continue to meet all inclusion and exclusion criteria. All screening procedures must be performed within 28 days of dose administration
* Female subjects of childbearing potential (defined as not surgically sterile or at least two years postmenopausal confirmed by a Screening Follicle Stimulating Hormone (FSH) level of > 40) must agree to use one of the following forms of contraception from 60 days prior through 90 days following the dose of Study Drug: hormonal (oral, transdermal, implant, or injection), barrier (condom, diaphragm with spermicide), intrauterine device (IUD), complete abstinence, or vasectomized partner (6 months minimum) or male subjects who are sexually active with women of child-bearing potential must agree to complete abstinence or to use a condom for 90 days following the dose of Study Drug;
* No clinically significant abnormal findings on physical examination, vital signs, ECG, or clinical laboratory evaluation during screening; and systolic blood pressure between 140 mm and 90 mm Hg and diastolic blood pressure between 90 mm and 45 mm Hg.
* Can understand and sign the informed consent document, can communicate with the investigator, and can understand and comply with the requirements of the protocol.

Exclusion Criteria:

* Have a past or present serious medical illness or other medical or social reason that in the opinion of the Principal Investigator, would jeopardize the safety of the subject or impact the validity of the study results;
* Participation in a clinical trial (other than a screening visit) within 60 days of study drug administration;
* Use of any over-the-counter or prescription medication within 14 days prior to the dose of Study Drug or during the study, with the exception of hormonal contraceptives for women of childbearing potential, unless approved by the Principal Investigator or use of beta-blockers within 30 days prior to dose of Study Drug or during the study;
* Donation of blood or plasma within 30 days of the dose of Study Drug and throughout the duration of the study and for male subjects, donation of sperm through the duration of the study;
* Women who are nursing, pregnant, suspected of being pregnant, or trying to become pregnant, or are lactating, have a positive serum pregnancy test at screening or urine pregnancy test prior to administration of Study Drug regardless of childbearing potential;
* Positive blood screen for HIV, hepatitis B surface antigen (HbSAg), or hepatitis C as Screening, or a positive urine screen for alcohol (Day -1 only) or, drugs of abuse, or cotinine at Screening and on Day -1;
* Have clinically significant abnormalities in laboratory values as judged by the clinical investigator;
* Have a history of alcoholism and/or drug abuse;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-02-17 (Actual); Study Completion 2019-02-17 (Actual)

PRIMARY OUTCOMES:
Safety of a single intravenous (IV) infusion of NPT189 (subjects experiencing adverse events) | Day 1 through to Day 49
  Summary of the frequency and percentage of

SECONDARY OUTCOMES:
Profile of pharmacokinetics (PK) of a single intravenous (IV) infusion of NPT189 (Cmax) | Day 1 through to Day 49
  Observed maximum concentration (Cmax)
Profile of pharmacokinetics (PK) of a single intravenous (IV) infusion of NPT189 (Tmax) | Day 1 through to Day 49
  Time of the maximum measured concentration (Tmax)
Profile of pharmacokinetics (PK) of a single intravenous (IV) infusion of NPT189 (AUClast) | Day 1 through to Day 49
  Area under the concentration-time curve from time zero to the last quantifiable concentration time-point (AUClast)
Profile of pharmacokinetics (PK) of a single intravenous (IV) infusion of NPT189 (AUCinf) | Day 1 through to Day 49
  Area under the concentration-time curve from time zero extrapolated to infinity (AUCinf)
Profile of pharmacokinetics (PK) of a single intravenous (IV) infusion of NPT189. Terminal elimination half-life (t 1/2) | Day 1 through to Day 49
  Terminal elimination half-life (t 1/2)
Profile of pharmacokinetics (PK) of a single intravenous (IV) infusion of NPT189. Clearance (CL) | Day 1 through to Day 49
  Clearance (CL)
Profile of pharmacokinetics (PK) of a single intravenous (IV) infusion of NPT189. Volume of distribution (Vd) | Day 1 through to Day 49
  Apparent volume of distribution (Vd)

CONTACTS AND LOCATIONS:
Overall Officials: Proclara Biosciences, Study Director — Proclara
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krishnan R, Tsubery H, Proschitsky MY, Asp E, Lulu M, Gilead S, Gartner M, Waltho JP, Davis PJ, Hounslow AM, Kirschner DA, Inouye H, Myszka DG, Wright J, Solomon B, Fisher RA. A bacteriophage capsid protein provides a general amyloid interaction motif (GAIM) that binds and remodels misfolded protein assemblies. J Mol Biol. 2014 Jun 26;426(13):2500-19. doi: 10.1016/j.jmb.2014.04.015. Epub 2014 Apr 22. PMID 24768993